CLINICAL TRIAL: NCT02830646
Title: Measurement of Kidney Function Indexed Extracellular Volume Before and After Obesity Surgery in Kidney Patients With Severe Obesity or Massive
Brief Title: Kidney Function Indexed Extracellular Volume Before and After Obesity Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14-AOI-09
Record Dates: First submitted 2015-05-12; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DFG mesure (Other): Measure the effect of gastric bypass on the report DFG / VEC
  Interventions: Other: DFG mesure

INTERVENTIONS:
Other: DFG mesure — Measure the effect of gastric bypass on the report DFG / VEC.

SUMMARY:
Obesity promotes chronic kidney disease and is accelerating its shift to the stage of renal replacement. Bariatric surgery is a treatment for severe or morbid obesity whose renal benefit is currently unknown. The glomerular filtration rate (GFR) is the best parameter to define the kidney function. It can be estimated using formulas by assaying endogenous markers (creatinine, cystatin C) or measured with an exogenous tracer glomerular filtration (51 Cr-EDTA).

Bariatric surgery alters the production of endogenous markers and the extracellular volume (VEC) with 2 important consequences on the assessment of GFR: the formula to estimate GFR is not possible to compare renal function before and after surgery because of the variation in production of endogenous glomerular filtration markers in the same subject; decreasing VEC predicted decreased GFR after surgery, since these parameters are in part proportional to each other.

Our working hypothesis is that bariatric surgery protects the kidneys of patients with chronic kidney disease. To demonstrate this, investigators propose to compare the ratio DFG / VEC before and after gastric bypass.

Goals The main objective is to measure the effect of gastric bypass on the report DFG / VEC. Secondary objectives are to assess the effect of gastric bypass on the albumin / urine creatinine and evaluate the performance of the main GFR estimating formulas in people with severe or morbid obesity.

ELIGIBILITY:
Inclusion Criteria:

* Topic GFR estimated by having the simplified formula of MDRD <60 ml / min / 1.73 m²
* Topic with BMI ≥ 40 kg / m², or ≥ 35 kg / m²
* Subject having at least one comorbidity could be improved after surgery after failure of medical treatment: hypertension , OSAHS and other severe respiratory disorders, severe metabolic disorders, particularly type 2 diabetes , debilitating musculoskeletal diseases, steatohepatitis nonalcoholic .
* Topic who signed the informed consent
* Topic affiliated to the social security
* Male or female Topics
* Elderly 18 to 70 inclusive

Exclusion Criteria:

* Non- Caucasian person because the necessary correction factors and not always available for the formula to estimate GFR ( Cockcroft , Salazar and Corcoran ) .
* No major under guardianship
* Nobody hospitalized without his consent and not protected by law
* Private person of liberty
* Pregnant Woman, knowing that a pregnancy test will be performed for women of childbearing age . Results will be communicated to the patient by a doctor of his choice.
* Rapidly progressive glomerulonephritis
* Nephrotic proteinuria ranking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ratio DFG / VEC | Month 12
  Average ratio DFG / VEC before and one year after gastric bypass

SECONDARY OUTCOMES:
Albumin / urine creatinine | Month 12
GFR estimation formula | Month 12
  GFR using the Cockcroft formulas , Salazar and Corcoran , simplified MDRD and CKD -EPI . Each of GFR estimation formula , we calculate the mean bias by the difference between the estimated value and the measured value and the percentage of patients with the value obtained by estimation is between -25 % and + 25 % in value measured ( awerage Within 50 or AW50 )

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France